CLINICAL TRIAL: NCT00302081
Title: Comparison of Three Regimens of PEG-Intron and Ribavirin in the Treatment of Chronic Hepatitis C, Genotype 2 or 3, in Previously Untreated Patients
Brief Title: Three Regimens of PegIntron Plus Ribavirin in Previously Untreated Chronic Hepatitis C, Genotype 2 or 3 (Study P03548)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03548
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Genotype 2 and Genotype 3
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG2b 1.5/R (24 weeks) (Active Comparator): PegIntron (peginterferon alfa-2b; SCH 54031) 1.5 mcg/kg QW SC plus ribavirin (SCH 18908) 800-1200 mg daily for 24 weeks
  Interventions: Biological: peginterferon alfa-2b (SCH 54031); Drug: ribavirin (SCH 18908)
- PEG 2b 1.0/R (24 weeks) (Experimental): PegIntron (peginterferon alfa-2b; SCH 54031) 1.0 mcg/kg QW SC plus ribavirin (SCH 18908) 800-1200 mg/day for 24 weeks
  Interventions: Biological: peginterferon alfa-2b (SCH 54031); Drug: ribavirin (SCH 18908)
- PEG2b 1.5/R (16 weeks) (Experimental): PegIntron (peginterferon alfa-2b; SCH 54031) 1.5 mcg/kg QW SC plus ribavirin (SCH 18908) 800-1200 mg/day for 16 weeks
  Interventions: Biological: peginterferon alfa-2b (SCH 54031); Drug: ribavirin (SCH 18908)

INTERVENTIONS:
Biological: peginterferon alfa-2b (SCH 54031) — 1.5 mcg/kg QW SC for 24 weeks
  Other Names: PegIntron (SCH 54031)
  Arms: PEG2b 1.5/R (24 weeks)
Biological: peginterferon alfa-2b (SCH 54031) — 1.0 mcg/kg QW SC for 24 weeks
  Other Names: PegIntron (SCH 54031)
  Arms: PEG 2b 1.0/R (24 weeks)
Biological: peginterferon alfa-2b (SCH 54031) — 1.5 mcg/kg QW SC for 16 weeks
  Other Names: PegIntron (SCH 54031)
  Arms: PEG2b 1.5/R (16 weeks)
Drug: ribavirin (SCH 18908) — 800-1200 mg daily for 24 weeks
  Other Names: REBETOL (SCH 18908)
  Arms: PEG 2b 1.0/R (24 weeks); PEG2b 1.5/R (24 weeks)
Drug: ribavirin (SCH 18908) — 800-1200 mg daily for 16 weeks
  Other Names: REBETOL (SCH 18908)
  Arms: PEG2b 1.5/R (16 weeks)

SUMMARY:
This is a randomized, open-label, multinational study designed to evaluate the "standard" regimen, PegIntron 1.5 µg/kg subcutaneously once weekly plus ribavirin 800-1200 mg daily [Arm PEG2b 1.5/R (24 weeks)], compared to a lower dose regimen, PegIntron 1.0 µg/kg subcutaneously once weekly plus ribavirin 800-1200 mg daily [Arm PEG2b 1.0/R (24 weeks)], using a 24 week treatment duration for both arms. Additionally, the study examined the efficacy of reduced treatment duration: PegIntron 1.5 µg/kg subcutaneously once weekly plus ribavirin 800-1200 mg for 16 weeks [Arm PEG2b 1.5/R (16 weeks)] .

DETAILED DESCRIPTION:
This is a randomized, open-label, multinational study designed to evaluate the "standard" regimen, PegIntron 1.5 µg/kg subcutaneously once weekly plus ribavirin 800-1200 mg daily [Arm PEG2b 1.5/R (24 weeks)], compared to a lower dose regimen, PegIntron 1.0 µg/kg subcutaneously once weekly plus ribavirin 800-1200 mg daily [Arm PEG2b 1.0/R (24 weeks)], using a 24 week treatment duration for both arms. Additionally, the study examined the efficacy of reduced treatment duration: PegIntron 1.5 µg/kg subcutaneously once weekly plus ribavirin 800-1200 mg for 16 weeks [Arm PEG2b 1.5/R (16 weeks)].

ELIGIBILITY:
Inclusion Criteria:

The subject must meet ALL of the criteria listed below for entry into the study:

* Hemoglobin >= 11 g/dL (females); >= 12 g/dL (males)
* Platelet count >= 100,000/mm^3
* Neutrophil count >= 1,500/mm^3
* Adult male or female chronic hepatitis C (CHC) patients (HCV-RNA-positive in serum) with compensated liver disease (Child-Pugh Score <7) and indication for treatment according on current consensus guidelines (1. NIH Consensus Conference on the Management of Hepatitis C, 2002; 2. German Consensus Conference on Hepatitis B and C, published in Z Gastro 2004; 42 (8): 677-730).
* >= 18 to =< 70 years of age
* At least one abnormal ALT value in the last year
* HCV genotype 2 or 3
* Not previously treated with any interferon or ribavirin alone or in combination
* TSH level must be within normal limits
* At the Screen Visit, glucose must be 70-140 mg/dL. Results between 116-140 mg/dL require repeat fasting glucose to be less than140 mg/dL and HbA1C less than or equal to 8.5%. HbA1C must be less than or equal to 8.5% in diabetic subjects (whether on medication or diet controlled).
* Female subjects cannot be pregnant or breastfeeding and must be either postmenopausal, surgically sterile or using 2 methods of birth control. While abstinence from sexual activity is the only certain method to prevent pregnancy, female patients of childbearing potential who are or who anticipate the possibility of becoming sexually active with a male partner must use a combination of the following 2 methods: (1)contraceptive pill or IUD or depot hormonal preparation (ring, injection implant); and (2) a barrier method of contraception such as diaphragm, sponge with spermicide, condom, or a method of birth control considered acceptable by the study physician. Contraceptive measures will be reviewed with female subjects at each visit. Dual methods of contraception must be used for 6 months after treatment discontinuation.
* Sexually active male subjects must be practicing acceptable methods of contraception (vasectomy, use of condom plus spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 7 months after stopping treatment
* Subjects must be willing to give written informed consent and able to adhere to dosing and visit schedules.
* Confirmation by the principal investigator or a sub-investigator that sexually active females of childbearing potential are practicing adequate contraception.
* A serum pregnancy test obtained at Screen Visit prior to the initiation of treatment must be negative
* Confirmation by the principal investigator or a sub-investigator that sexually active male subjects are practicing a method of contraception considered acceptable (vasectomy, condom plus spermicide, plus relationship with a female partner who practices an acceptable method of contraception). Contraception must be used during the treatment period and for seven months (or 6 months, according to local label) after the completion of therapy, including condom use by male subjects with pregnant partners.
* For subjects with a history of hypertension or diabetes, written clearance from an ophthalmologist has to be obtained prior to treatment start

Exclusion Criteria:

* Patients younger than 18 years
* Patients older than 70 years of age.
* Positive Anti-HIV antibodies
* Positive HBsAg antibodies
* Patients with severe renal dysfunction or creatinine clearance < 50 mL/min must not be treated with PEG-Intron -Rebetol
* Pregnant women, women who plan to become pregnant, male subjects whose partner wants to become pregnant, and breastfeeding women.
* Suspected hypersensitivity to any interferon or ribavirin product.
* Subject has used any investigational product within 30 days prior to enrollment
* Subject is participating in any other clinical study
* Any cause of liver disease other than chronic hepatitis C, including but not limited to:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Non-alcoholic steatohepatitis (NASH)
  * Drug-related liver disease
* Active malignant disease or suspicion or history of malignant disease within five previous years (except for adequately treated basal cell carcinoma)
* Known coagulation diseases such as hemophilia; hemoglobin diseases (e.g. thalassemia)
* Known G6PD deficiency
* Evidence of advanced liver disease such as history or presence of ascites, bleeding varices, or hepatic encephalopathy.
* Subjects with organ transplants, except for corneal or hair transplant.
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of study, such as:

  * Preexisting psychiatric condition, especially moderate to severe depression, or a history of severe psychiatric disorder, such as psychosis, suicidal ideation, or suicide attempts. Severe depression includes the following: hospitalization for depression; electroconvulsive therapy for depression; or depression causing a prolonged absence from work or significantly altering daily functions. Subjects with mild depression may be considered for entry into the study provided that a pre-treatment assessment demonstrates that the subject's emotional status is clinically stable, in which case a management plan must be formulated for the subject; this management plan will become a part of the subject's medical record.
  * Craniocerebral trauma which is not a concussion or active seizure disorders requiring medication.
  * Clinically significant ECG abnormalities and/or cardiovascular dysfunction within 6 previous months (e.g., angina, congestive heart failure, recent myocardial infarction, or significant arrhythmia).
  * Chronic lung disease (e.g., chronic obstructive lung disease)
  * Poorly controlled diabetes mellitus
  * Immune-mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis)
  * Clinical gout
* Subject is or was a substance abuser, such as alcohol (80 gm/day or more), methadone, IV, oral or inhaled drugs. To be considered for inclusion into the protocol, the subject must have abstained and agree to abstain from using any of the above for at least 6 months. Subjects treated with buprenorphine (Subutex) who have been stable for 6 months may be included
* Any other condition that, in the investigator's opinion, could determine that subject's participation in the study is not indicated or could interfere with the subject's participation in and completion of study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2003-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Manns M, Zeuzem S, Sood A, Lurie Y, Cornberg M, Klinker H, Buggisch P, Rossle M, Hinrichsen H, Merican I, Ilan Y, Mauss S, Abu-Mouch S, Horban A, Muller TH, Welsch C, Chen R, Faruqi R, Pedicone LD, Wedemeyer H. Reduced dose and duration of peginterferon alfa-2b and weight-based ribavirin in patients with genotype 2 and 3 chronic hepatitis C. J Hepatol. 2011 Sep;55(3):554-563. doi: 10.1016/j.jhep.2010.12.024. Epub 2011 Jan 13. PMID 21237227

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 696 subjects were randomized. 14 subjects never received any study drug and, therefore, were excluded from the Intent to Treat (ITT) population. ITT population consisted of 682 subjects.
Groups:
- PEG2b 1.0/R (24 Weeks): PegIntron (peginterferon alfa-2b; SCH 54031) 1.0 mcg/kg QW SC plus ribavirin (SCH 18908) 800-1200 mg/day for 24 weeks
Period: Overall Study
Arm/Group | PEG2b 1.5/R (24 Weeks) | PEG2b 1.0/R (24 Weeks) | PEG2b 1.5/R (16 Weeks)
Started | 237 | 229 | 230
Completed | 181 | 186 | 178
Not Completed | 56 | 43 | 52
Not completed — Adverse Event | 6 | 5 | 4
Not completed — Lost to Follow-up | 21 | 18 | 28
Not completed — Withdrawal by Subject | 8 | 12 | 8
Not completed — Protocol Violation | 5 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 5
Not completed — Death | 2 | 1 | 0
Not completed — Other | 13 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG2b 1.5/R (24 Weeks) | PEG2b 1.0/R (24 Weeks) | PEG2b 1.5/R (16 Weeks) | Total
Number analyzed (Participants) | 230 | 224 | 228 | 682
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (10.2) | 39.9 (11.2) | 39.7 (11.1) | 39.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 78 | 80 | 249
  Male | 139 | 146 | 148 | 433

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Achieve a Sustained Virologic Response (SVR)
Description: A sustained virologic response is defined as undetectable hepatitis C virus ribonucleic acid [HCV-RNA] 24 weeks post-treatment. Serum HCV-RNA is measured by HCV-PCR in local laboratories. HCV-RNA below the limit of detection is considered undetectable.
Time Frame: 24-week treatment duration for Arms [Peg2b 1.5/R(24 weeks)] and [PEG2b 1.0/R(24 weeks]); 16-week treatment duration for Arm [PEG2b 1.5/R(16 weeks]. Follow-up of 24 weeks for each arm.
Population: Intent-to-Treat (ITT) population
Measure: Number; unit: participants
Arm/Group | PEG2b 1.5/R (24 Weeks) | PEG2b 1.0/R (24 Weeks) | PEG2b 1.5/R (16 Weeks)
Number analyzed (Participants) | 230 | 224 | 228
participants | 153 | 144 | 129
Statistical Analysis 1: Comparison: PEG2b 1.5/R (24 Weeks) vs PEG2b 1.0/R (24 Weeks); This is an evaluation of the effect of the peginterferon alfa-2b dose (1.0 vs 1.5 micrograms/kg/week) on the primary outcome measure; Test type: Non-Inferiority or Equivalence — Noninferiority for SVR was concluded if the lower limit of the one-sided 95% CI was greater than -10%. Otherwise, noninferiority was concluded for both dose and treatment duration comparisons if the lower limits of the two-sided 95% CIs were greater than -10%; p = 0.041, z-test (non-inferiority margin=-0.1) — The Hochberg procedure was used to adjust for the multiple comparisons ([PEG2b 1.0/R(24 weeks)] - [PEG2b 1.5/R(24 weeks]) and ([PEG2b 1.5/R(16 weeks)]-[PEG2b 1.5/R(24 weeks)]); SVR rates are 0.665 (153/230 subjects) in the 1.5-dose group and 0.643 (144/224 subjects) in the 1.0-dose group, for a risk difference of -0.02; Risk Difference (RD) = -0.02, 95% CI [-0.10 to 1]
Statistical Analysis 2: Comparison: PEG2b 1.5/R (24 Weeks) vs PEG2b 1.5/R (16 Weeks); This is an evaluation of the effect of treatment duration (24 weeks vs 16 weeks) on the primary outcome measure; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.495, z-test (non-inferiority margin=-0.1) — The Hochberg procedure was used to adjust for the multiple comparisons ([PEG2b 1.0/R(24 weeks)] - [PEG2b 1.5/R(24 weeks]) and ([PEG2b 1.5/R(16 weeks]-[PEG2b 1.5/R(24 weeks]); SVR rates are 0.665 (153/230 subjects) in the 24-week group and 0.566 (129/228 subjects) in the 16-week group, for a risk difference of -0.10; Risk Difference (RD) = -0.10, 95% CI [-0.17 to 1]

2. Secondary Outcome: Virologic Response Rates at the End of Therapy. Biochemical Responses as Determined by ALT and AST Levels at the End of Treatment and at the End of Follow up.
Description: Virologic response is defined as undetectable hepatitis C virus ribonucleic acid (HCV-RNA) in the serum. A blood test is used to measure the level of ALT and AST. ALT response was defined as ALT<40 IU/L (international units per liter).
  This was not a prespecified key secondary outcome.
Time Frame: End of treatment: 24 weeks for arms [PEG2b 1.5/R (24 weeks)] and [PEG2b 1.0/R (24 weeks)]; 16 weeks for arm [PEG2b 1.5/R (16 weeks)]. Follow-up of 24 weeks for each arm.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | PEG2b 1.5/R*(24 Weeks) | PEG2b 1.0/R*(24 Weeks) | PEG2b 1.5/R*(16 Weeks)
Serious Adverse Events (participants affected / at risk) | 14/230 | 11/224 | 7/228
Other Adverse Events (participants affected / at risk) | 196/230 | 187/224 | 201/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG2b 1.5/R*(24 Weeks) (N=230) | PEG2b 1.0/R*(24 Weeks) (N=224) | PEG2b 1.5/R*(16 Weeks) (N=228)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
AMAUROSIS FUGAX (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
VISUAL DISTURBANCE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
HERNIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
COMA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
AGGRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ANGER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
NERVOUSNESS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PERSECUTORY DELUSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PREGNANCY OF PARTNER (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG2b 1.5/R*(24 Weeks) (N=230) | PEG2b 1.0/R*(24 Weeks) (N=224) | PEG2b 1.5/R*(16 Weeks) (N=228)
ANAEMIA (Blood and lymphatic system disorders) | 22 (27) | 11 (12) | 25 (26)
LEUKOPENIA (Blood and lymphatic system disorders) | 14 (16) | 17 (18) | 22 (22)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 11 (11) | 11 (14) | 12 (12)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 11 (11) | 18 (21) | 9 (13)
DIARRHOEA (Gastrointestinal disorders) | 22 (28) | 27 (28) | 16 (18)
DRY MOUTH (Gastrointestinal disorders) | 12 (12) | 5 (5) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 11 (13) | 20 (25) | 14 (18)
NAUSEA (Gastrointestinal disorders) | 27 (32) | 26 (29) | 31 (34)
VOMITING (Gastrointestinal disorders) | 6 (6) | 12 (13) | 7 (7)
ASTHENIA (General disorders) | 44 (74) | 62 (75) | 45 (63)
CHILLS (General disorders) | 13 (15) | 13 (14) | 16 (17)
FATIGUE (General disorders) | 52 (64) | 50 (57) | 36 (43)
INFLUENZA LIKE ILLNESS (General disorders) | 29 (35) | 21 (24) | 23 (31)
INJECTION SITE ERYTHEMA (General disorders) | 26 (27) | 31 (40) | 17 (18)
IRRITABILITY (General disorders) | 8 (11) | 14 (15) | 10 (10)
PAIN (General disorders) | 17 (56) | 13 (55) | 13 (53)
PYREXIA (General disorders) | 87 (328) | 83 (300) | 101 (296)
HAEMOGLOBIN DECREASED (Investigations) | 12 (14) | 7 (7) | 11 (14)
WEIGHT DECREASED (Investigations) | 29 (29) | 24 (24) | 31 (31)
ANOREXIA (Metabolism and nutrition disorders) | 28 (32) | 11 (12) | 22 (23)
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 (8) | 14 (14) | 12 (13)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 25 (27) | 17 (22) | 24 (27)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (14) | 11 (12) | 12 (12)
MYALGIA (Musculoskeletal and connective tissue disorders) | 35 (64) | 27 (31) | 34 (35)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (12) | 16 (22) | 15 (16)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 9 (9) | 13 (13) | 2 (2)
DIZZINESS (Nervous system disorders) | 13 (16) | 5 (7) | 9 (10)
HEADACHE (Nervous system disorders) | 52 (74) | 57 (98) | 58 (78)
DEPRESSED MOOD (Psychiatric disorders) | 25 (26) | 16 (17) | 19 (19)
DEPRESSION (Psychiatric disorders) | 19 (20) | 11 (13) | 7 (7)
INSOMNIA (Psychiatric disorders) | 17 (19) | 11 (11) | 10 (11)
SLEEP DISORDER (Psychiatric disorders) | 19 (22) | 6 (6) | 7 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 22 (28) | 22 (23)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 14 (15) | 9 (9)
ALOPECIA (Skin and subcutaneous tissue disorders) | 48 (49) | 36 (37) | 31 (31)
DRY SKIN (Skin and subcutaneous tissue disorders) | 13 (14) | 25 (26) | 15 (16)
PRURITUS (Skin and subcutaneous tissue disorders) | 29 (35) | 44 (49) | 23 (25)
RASH (Skin and subcutaneous tissue disorders) | 14 (15) | 15 (18) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less